CLINICAL TRIAL: NCT07072169
Title: A Clinical Study to Investigate Safety, Tolerability, and Preliminary Efficacy of mRNA Encoding CD19/CD3 T Cell Engager (ABO2203) in Adult Patients With Relapsed or Refractory B-NHL
Brief Title: A Study of mRNA Encoding CD19/CD3 T Cell Engager (ABO2203) in Patients With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma (B-NHL)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABO2203-003
Record Dates: First submitted 2025-05-26; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-05

CONDITIONS: B-cell Non-Hodgkin Lymphoma
Keywords: mRNA, CD19/CD3, T cell engager, B-NHL
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A study of mRNA encoding CD19/CD3 T cell engager (ABO2203) in patients with relapsed or refractory B (Experimental): ABO2203
  Interventions: Drug: ABO2203 Injection

INTERVENTIONS:
Drug: ABO2203 Injection — SC or IV

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, as well as preliminary efficacy of mRNA encoding CD19/CD3 T cell engager (ABO2203) in adult patients with relapsed or refractory CD19-positive B-NHL, This study included dose escalation and dose expansion parts.

ELIGIBILITY:
Key-Inclusion Criteria:

* ≥18 years and ≤75 years of age at time of informed consent
* Participants with histologically and/or cytologically confirmed relapsed or refractory CD19-positive B-cell non-Hodgkin lymphoma
* With at least one of evaluable/measurable target lesions per Lugano 2014 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2
* Life expectancy of ≥3 months
* Sufficient organ function

Key-Exclusion Criteria:

* Central nervous system lymphoma
* Previously undergone allogeneic hematopoietic stem cell transplantation or other organ transplants
* Any other prior malignancy active within the previous 5 years, except for skin basal cell cancer that has been cured, or carcinoma in situ of the cervix
* History of active autoimmune diseases
* History of interstitial lung disease, tuberculosis, or other diseases that affect pulmonary function in the past or currently
* Uncontrolled disease, including but not limited to uncontrolled diabetes, hypertension, active infections, active peptic ulcers, thromboembolic disease requiring anticoagulation, etc.
* Severe cardiovascular diseases
* History of severe allergies to protein-based drugs or any component of the study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
A study of mRNA encoding CD19/CD3 T cell engager (ABO2203) in patients with relapsed or refractory B-cell non-Hodgkin lymphoma (B-NHL) | From the first dose to 30 days after the last dose of ABO2203 treatment
  The incidence and severity of adverse events evaluated by Common Terminology Criteria for Adverse Events (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Wei li Zhao, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China